CLINICAL TRIAL: NCT06027931
Title: 12-months Clinical and Radiographical Outcomes of Root Canal Treatment After Traditional Versus Conservative Access Cavities: A Randomized Controlled Clinical Trial
Brief Title: Traditional Versus Conservative Access Cavities Cleaning Ability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Alani, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahmed Alani 1983
Record Dates: First submitted 2023-03-28; First posted 2023-09-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Root Canal Infection; Root Canal Treatment
Keywords: Root Canal,CFU

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Access Opening (Experimental): Root canal treatment using Conservative Access Opening type.
  Interventions: Procedure: Conservative Access Opening, Traditional Access Opening
- Traditional Access Opening (Experimental): Root canal treatment using Traditional Access Opening type.
  Interventions: Procedure: Conservative Access Opening, Traditional Access Opening

INTERVENTIONS:
Procedure: Conservative Access Opening, Traditional Access Opening — Conservative Access Opening will be used and evaluated for cleaning ability versus Traditional Access Opening.

SUMMARY:
Aims of the study:

1. Assess the clinical and radiographical outcomes (success/failure) of root canal treatments performed after traditional vs conservative access cavities in permanent posterior teeth after one-year follow-up.
2. Assess the level of disinfection in root canals accessed by traditional vs conservative access cavities in permanent posterior teeth before obturation.

Null hypothesis:

1. There is no difference in the clinical and radiographical outcomes of root canal treatments performed after traditional and conservative access cavities preparation in posterior teeth after one-year of follow-up.

DETAILED DESCRIPTION:
Objectives:

1- Primary outcomes:

1. A single-blind, 2- arms, parallel 2-groups, randomized controlled clinical trial will be conducted in two groups of patients to assess the clinical and radiographical outcomes (success/failure) of root canal treatments after one year follow-up of posterior teeth accessed by traditional or conservative access cavities using CBCT as a strict radiographic adjunct in the assessment in addition to the conventional clinical tests and the 2- dimensional radiographs.

   The successful outcome will include:

   I. The absence of clinical signs and symptoms (pain, tenderness to percussion, sinus tract, swelling).

   II. No pathosis is evident on the recall CBCT such as root resorption, new furcal, or periapical rarefaction.

   III. Complete radiographic healing or reduction in the radiolucency if periapical rarefaction was present preoperatively.

   The clinical assessment will be performed by a blind clinical observer and the radiographical outcome will include an assessment of pretreatment and posttreatment CBCT scans by blinded two observers (a consensus panel).
2. A microbiological study will be performed to assess the level of disinfection in the root canals accessed by traditional versus the conservative access cavities by measuring the total bacterial count before and after the instrumentation of the root canals.

   2- Secondary outcomes of the trial:

   1- Assessment of crown fracture during the one-year follow-up period (if any). 2- Assessment of fracture file events during treatment phase. 3- Assess the accuracy of CBCT vs periapical radiographs in detection of periapical lesion in baseline and follow-up radiographical assessment.

   Materials & Method:

   Study design:

   This single blind, 2-arms, parallel groups, randomized clinical trial study is planned to be conducted in a private dental center in Baghdad, Iraq. Ethical approval will be granted from the Ethics committee in the College of Dentistry/University of Baghdad.

   CBCT scan and periapical radiograph will be taken for each case preoperatively, and another CBCT will be acquired after 1-year follow-up. These scans and radiographs will be assessed by a consensus panel of two academic endodontists in the department of Esthetic and restorative dentistry.

   A customized case sheet was prepared to be filled before starting with the treatment, after getting patient approval on participation in the study and signature the consent form. Case sheets and consent forms in Arabic and English languages are in the last pages in this protocol.

   3.2. Sample size calculation: This study was designed to have 80% power with an alpha margin of error of 5%, the sample size was calculated using G-power to detect an expected difference of 25% in failed outcomes between the two groups after one year of follow-up, a total sample size of 84 root canal treatments in two groups (each group = 42) was calculated anticipating 10% loss of follow-up after one year.

   Cases selection:

   Inclusion criteria: mature maxillary and mandibular (first molars, first, and second premolars) that have clinical signs and symptoms of irreversible pulpitis or necrotic pulps that may or may not show apical periodontitis or chronic apical lesions on the preoperative CBCT scan or periapical radiograph.

   Exclusion criteria: pregnancy, immunosuppression, patients received radiotherapy, unrestorable teeth, teeth with periodontal probing depths greater than 3 mm, uncontrolled periodontal disease, presence of airways disease or allergy, vertical root fractures, signs of root resorption, or patient age over 70 years old.

   3.4. Randomization and patients Grouping: Block randomization will be performed using computer software, the tooth will be the unit of randomization. The following factors will be equalized during the allocation of teeth to the study arms: Gender (male/female), Age median, tooth type (molar/premolar), periapical lesion (presence/absence).

   Materials and Equipment:

   List of materials:

   1. Barbed broaches (Dentsply Maillefer, USA). 2. Disposable nitril gloves (Provi, Malaysia). 3. Disposable syringe 5ml (Malaysia) 4. EDTA solution 17% (Produits Dentaires SA, Switzerland) 5. Glyde (Dentsply, Sirona). 6. Bioceramic root canal sealer (BioRoot ™Flow, Septodont). 7. K-files #10 (Dentsply Maillefer, Switzerland). 8. K-files #15 (Dentsply Maillefer, Switzerland). 9. NAOCL 5.25 % (Cerkamed, Poland). 10. Protaper Gold rotary files (Dentsply, Sirona). 11. Transfer sponges (Dentsply Maillefer, Switzerland). 12. Irrigation needles 0.3 x 25(Cerkamed, Poland). 13. Normal saline. 14. Paper point (Dentsply, Maillefer, Switzerland). 15. Dam sheets (Sanctuary). 16. Gutta percha cones (Dentsply Maillefer, Switzerland). 17. Burs (Endo Z).

   Instruments:
   1. Diagnostic instruments (mirror, probe, and Tweezers) (Medesey, Italy).
   2. Rubber Dam kit.
   3. Endodontic plugger (Medesey, Italy)
   4. Endodontic ruler (Dentsply, Sirona).
   5. Ultrasonic Endotips.
   6. Ethyl chloride and electric pulp tester.

   Equipment:
   1. X-Smart IQ Cordless Endodontic Motor (Dentsply, Sirona).
   2. High-speed handpiece (Bien Air, Optima, Switzerland).
   3. Low-speed handpiece (NSK, Japan)
   4. Apex locator (NSK, Apex II, Japan).
   5. An ultrasonic scaler (Ultramint & Ultramint Pro, Eighteeth).

   Endodontic procedure:

   1. Tooth Preparation: An individual patient's data, including case history, clinical and radiological assessment, treatment plan and periodic follow-up of the patients will be recorded. Preoperative CBCT and periapical radiograph will be taken for each patient before starting the treatment. The time required for complete endodontic procedure will be recorded from the start of treatment for each case. Following anesthesia caries removal will be performed and restorability will be confirmed. In case of missing walls (Class II) cavity, pre-endodontic build-up will be performed. With rubber dam isolation, endodontic treatment will be started, after a straight-line access cavity is prepared by maintaining standard protocol, with confirmation of patency with size 8 and 10 k files. Working length will be confirmed with an electronic apex locator and radiograph, canals will be enlarged using Protaper Gold file system to Size F2 at minimum and for MB2 size F2 will be considered the master apical file with 2% sodium hypochlorite irrigation throughout the procedure, finally, the irrigant will be left in the canal and activated by smooth ultrasonic file (size 15, 0.02 taper) that placed into the canal to 1 mm short of the WL without touching the walls, enabling it to vibrate freely for 1 min (Hegde and Arora, 2015). Then final irrigation was done with 17% liquid ethylenediamine tetra acetic acid (17%EDTA) to remove the smear layer then irrigation with 2.5% NaOCl solution was placed and agitated for 60 seconds followed by a final irrigation with 1 mL of saline solution (Tavares, 2020). The canals will be dried with paper point, and master cone (gutta-percha) to be selected depending on master apical file for canals. Obturation will be performed with bioceramic sealer (BC) using single cone technique.

   2 Bacterial Count (Sample Collection): During sample collection, a sterile absorbent paper points size F2 will be introduced individually in the pulp chamber space before access cavity preparation and remained in this position for 60 seconds. After this, the paper point will be stored in a sterile microtube (2 mL) containing 1 mL pyrogenic water for subsequent microbiological analysis of Colony Forming Unit (CFU). This will be considered the base line measurement. After access cavity preparation and instrumentation, the second paper point will be inserted in the root canal space and remain in this position for 60 seconds and then will be stored in a sterile microtube (2 mL) containing 1 mL pyrogenic water for subsequent microbiological analysis of Colony Forming Unit (CFU). This will be regarded as a second measurement for comparison purposes.

   3. Obturation BC sealer is chosen to be used in this study as it has exceptional dimensional stability and does not shrink upon setting; it is non-resorbable inside root canal. Furthermore, the formation of calcium hydroxide as a by-product of the setting reaction (initiated by moisture present in dentinal tubules) produces a very high alkaline pH (12.8) rendering the material antibacterial. It exhibits excellent biocompatibility; significant stimulation of periodontal regeneration and it is osteoconductive. All teeth will be referred back for final restoration within 1 month.

   Bioceramic root canal sealer is supplied in premix tube with disposable tips of narrow caliber. The syringe cap is to be removed from the syringe and intra canal tip to be attached with a clockwise twist to the hub of the syringe. Sealer will be injected into the coronal half of the canal and premeasured master gutta-percha (GP) point will be inserted it into the canal very slowly. GP carried sufficient sealer to the apex. Excess GP points will be removed from the pulp chamber by a heated plugger.

   4. Review of patients: Patients will be reviewed with a clinical and radiographic examination, one year after treatment. During this examination, CBCT will be taken using the same exposure settings as the initial scan.

   5. Radiographic assessment: Two examiners who had not been involved in clinical examination or treatment of patients will assess all the CBCT scans. Preoperative and follow-up CBCT images will be assessed for the presence of apical periodontitis, and dimension of periapical lesion.

   The assessment will be carried out on the coronal and sagittal slices at the equatorial level of the tooth of interest.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of root canal disease.
* Must be able to undergo endodontic treatment.

Exclusion Criteria:

* pregnancy patients.
* patients received radiotherapy.
* patient age over 70 years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-05-12 (Estimated); Study Completion 2024-05-12 (Estimated)

PRIMARY OUTCOMES:
The absence of clinical signs and symptoms in participants. | 1 year
  (pain, tenderness to percussion, sinus tract, swelling).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Ali, Ph.D, Study Director — University of Baghdad
Locations (1):
- Private Dental Center, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
CBCTs